CLINICAL TRIAL: NCT05269160
Title: A Phase I/II Study of Dermaprazole for Radiation Dermatitis in Post-Mastectomy Breast Cancer Patients.
Brief Title: Topical Dermaprazole for Radiation Dermatitis in Breast Cancer Patients (TOPAZ)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michelle S Ludwig (Other)
Responsible Party: Sponsor-Investigator, Michelle S Ludwig, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: H-45698
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Radiation Dermatitis; Breast Cancer
Keywords: Radiation dermatitis; post-mastectomy; radiation therapy; breast cancer
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dermaprazole 1% (Breast) (Experimental): Dermaprazole cream at a concentration of 1% will be applied to the skin twice daily starting from CT simulation throughout the radiation treatment period.
  Interventions: Drug: Dermaprazole 1%
- Dermaprazole 2% (Breast) (Experimental): Dermaprazole cream at a concentration of 2% will be applied to the skin twice daily starting from CT simulation throughout the radiation treatment period.
  Interventions: Drug: Dermaprazole 2%

INTERVENTIONS:
Drug: Dermaprazole 1% — Dermaprazole cream at a concentration of 1% will be applied to the irradiated area twice daily for up to 7 weeks
  Arms: Dermaprazole 1% (Breast)
Drug: Dermaprazole 2% — Dermaprazole cream at a concentration of 2% will be applied to the irradiated area twice daily for up to 7 weeks
  Arms: Dermaprazole 2% (Breast)

SUMMARY:
Radiotherapy is a mainstay of treatment in breast cancer treatment, in the adjuvant setting. Radiation dermatitis occurs in up to 65% of these patients; currently, there is no standard of care for this treatment-related toxicity. The aim of this study is to investigate the safety and tolerability (Phase I) and preliminary efficacy (Phase II) of prophylactic esomeprazole cream (termed "Dermaprazole") in patients who require radiation for breast cancer in the adjuvant setting.

DETAILED DESCRIPTION:
All study participants will begin using Dermaprazole for 1-2 weeks prior to receiving radiation. During the CT Simulation, study participants will be instructed to apply Dermaprazole in a "patch test" area - an area of the chest outside of the field of radiation. This is to assess for immediate skin reactions including itching, irritation and allergy. If there are no immediate allergic reactions at the conclusion of the simulation visit, the study participant will be instructed to apply the cream in the patch test for 2-4 days to assess for contact dermatitis and if no itching or rash at that time (evaluation will be conducted via phone call). Patients will be questioned regarding any visible skin changes or irritation (itching, peeling, scaling), and patients responding in the affirmative will be asked to present for clinic visit or send photographs for visual classification according to the scale outlines in Table 1 below. Skin reactions matching a score of 3 will be evaluated with a second clinic visit between 2 to 7 days after initial application. Any skin reactions of score 4 or 5 at final assessment will be deemed to be positive for allergic contact dermatitis, and patients will be deemed positive for allergic contact dermatitis.

Two dose levels of Dermaprazole (1% and 2%) will be evaluated in the combination Phase I/II dose escalation/de-escalation BOIN design study evaluating preliminary efficacy at the Maximum Feasible Dose (MFD). The Dermaprazole will be initiated at a dose of 1% and escalated to 2% as appropriate based on the number of adverse events. A Dose Limiting Toxicity (DLT) will be defined as any of the following: a) any > Grade 2 skin toxicity outside the radiation field (Macules/ papules covering 10-30% of the area with or without symptoms of pruritus, burning, tightness), b) any > Grade 2 radiation dermatitis (Moderate to brisk erythema; patchy moist desquamation, within the radiation field that is probably or definitely related to Dermaprazole. Dermatitis will be evaluated by a radiation oncologist on a weekly basis using the Common Terminology Criteria for Adverse Events (CTCAE) V5.0 criteria. Patient reported quality of life will be evaluated using a validated survey instrument called SkinDex16.

ELIGIBILITY:
Inclusion Criteria:

1. Women with breast cancer, treated with ipsilateral i) Simple (total) mastectomy, OR ii) Modified radical mastectomy, OR iii)Radical mastectomy, OR iv) Segmental mastectomy, OR v) Skin sparing/nipple sparing mastectomy
2. Histological diagnosis of invasive ductal or lobular carcinoma (diagnosed within 2 years of enrollment)
3. Planned to receive adjuvant chest wall radiation of at least 40Gy or higher biologically equivalent dose (BED)
4. Age 18 years or older
5. Women of childbearing potential (any woman with menses in the last 12 months) must agree to pregnancy testing and contraceptive use throughout the study period. Testing consists of human chorionic gonadotropin (HCG) urine testing, which if suspected to be falsely positive may be confirmed by ultrasound. If ultrasound is negative, patient is considered not pregnant and eligible for inclusion in the study. In addition to routine contraception method such as barrier devices, hormonal methods, and intrauterine devices, heterosexual celibacy, and surgical sterility (hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or a partner with history of vasectomy) is considered acceptable. If a celibate patient chooses to become sexually active during the study period, she must use one of the listed methods of contraception throughout the study period.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
7. Written Informed Consent
8. History and Physical within 12 weeks of enrollment

Exclusion Criteria:

1. Prior chest wall radiotherapy
2. Any serious medical condition or illness that would preclude the safe administration of the study drug including, but not limited to: active infection, symptomatic heart failure, unstable angina, psychiatric illness or social situations that would limit compliance with treatment
3. Concurrent chemotherapy
4. Biopsy-proven epidermal involvement or positive margins
5. Open wound at time of consultation, or delayed surgical wound healing as defined as open wound >8 weeks post-op
6. Known active collagen vascular disease such as systemic lupus erythematous, scleroderma or dermatomyositis.
7. Allergy or sensitivity to proton pump inhibitors
8. Pregnancy or breast feeding
9. Use of clopidrogrel, St. Johns Wort, rifampin, or methotrexate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-Limiting Toxicity(DLT) in phase I | from the first day applying the Dermaprazole cream until 1 month after the subject has completed their last radiation treatment
  A DLT is defined as any of the following:1) Any > Grade 2 skin toxicity outside the radiation field (Macules/ papules covering 10-30% of the area with or without symptoms of pruritus, burning, tightness); 2). Any > Grade 2 radiation dermatitis (Moderate to brisk erythema; patchy moist desquamation, mostly confined to skin folds and creases; moderate edema) within the treatment field that is probably or definitely related to Dermaprazole. Dermatitis will be evaluated by a radiation oncologist on a weekly basis using the Common Terminology Criteria for Adverse Events (CTCAE) V5.0 criteria. Patient reported quality of life will be evaluated using a validated survey instrument called SkinDex16.
Rate of clinically bothersome radiation dermatitis at maximum feasible dose in phase II | at weekly during radiation treatment, up to 7 weeks
  Radiation dermatitis will be determined by the radiation oncologist and defined using NCI Common Terminology Criteria for Adverse Events (CTCAE version 5) for dermatitis radiation. In particular, the individual components of radiation dermatitis will be recorded: erythema, desquamation, edema, bleeding, skin necrosis and skin ulceration.

SECONDARY OUTCOMES:
Rate of grade 2 or higher acute radiation dermatitis | from the first day the subject applies the cream to the end of the 6 month follow up period
  The proportion of patients with maximum observed acute grade 2, 3, and 4 skin reactions will be expressed in percentage. In particular, the individual components of radiation dermatitis will be recorded: erythema, desquamation, edema, bleeding, skin necrosis and skin ulceration.
Median- occurrence time of grade 2 or higher acute radiation dermatitis | from the first day the subject applies the cream to the end of the 6 month follow up period
  Median-occurrence of grade 2 or higher acute radiation dermatitis time on the Kaplan-Meier method is defined as the time between the first time of applying the cream and the time of occurrence of grade 2 or higher acute radiation dermatitis.
Median-healing time of grade 2 or higher acute radiation dermatitis develops | from the first day the subject applies the cream to the end of the 6 month follow up period
  Median-healing time of grade 2 or higher acute radiation dermatitis developing time on the Kaplan-Meier method is defined from time to develop the grade 2 or higher acute radiation dermatitis after applying the cream to healing the event.
Median of the peak score of each QOL component | at before and after Dermaprazole cream application at the CT simulation visit, weekly during radiation treatment up to 7 weeks, 1 and 6 month follow-up after completion of all radiation therapy
  Patient reported quality of life will be evaluated using a validated survey instrument called SkinDex16 questionnaire for QOL. The Skindex-16 assessment tool is designed to capture patient-reported assessments of subjective adverse effects. It consists of a short 16-item assessment completed by the patient, with each item rated on a 7-point Likert scale (0=never bothered to 6=always bothered).
Number of missed treatments due to skin toxicity | at weekly during radiation treatment, up to 7 weeks
  The missing numbers of treatment due to skin toxicity will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Ludwig, MD, MPH, PhD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine Medical Center - McNair Campus, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas